CLINICAL TRIAL: NCT05392894
Title: A Multi-centre Open Randomised Controlled Trial to Assess the Effect of Related Haplo-donor Haematopoietic Stem Cell Transplantation Versus Standard of Care (no Transplant) on Treatment Failure at 24 Month in Adults With Severe Sickle Cell Disease
Brief Title: RElated Haplo-DonoR Haematopoietic stEm Cell Transplantation for Adults With Severe Sickle Cell Disease
Acronym: REDRESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); University of Sheffield (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University College London Hospitals (Other); Manchester University NHS Foundation Trust (Other Government); St George's University Hospitals NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS: 312212
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle; Haploidentical; Stem cell; Transplant
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): The comparator arm is standard medical care for this patient population. Standard medical care may include all currently available non-trial therapies for SCD.
  Interventions: Other: Standard medical care
- Haploidentical stem cell transplantation (Experimental): Participants receiving Haploidentical Stem Cell Transplantation will receive the transplant conditioning regimen as per the standard transplant protocol. Stem cells from a haploidentical donor will be infused on Day 0 according to standard institutional practices. Bone marrow is the preferred stem cell source however peripheral blood may be used as an alternative where required due to donor reasons.
  Interventions: Procedure: Haploidentical stem cell transplantation

INTERVENTIONS:
Procedure: Haploidentical stem cell transplantation — Stem cell transplant from bone marrow or peripheral blood from haploidentical donor using standard nationally approved transplant procedure.
  Arms: Haploidentical stem cell transplantation
Other: Standard medical care — Standard medical care may include any currently available therapies for SCD patients. These may or may not include regular elective transfusion therapy or medications such as hydroxycarbamide.
  Arms: Standard of care

SUMMARY:
The purpose of this clinical trial is to evaluate the clinical and cost effectiveness of Haploidentical Stem Cell Transplantation (SCT) for adults with severe sickle cell disease (SCD), who have failed other therapies or are intolerant of existing therapies or require chronic transfusions to prevent on-going complications of SCD.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age ≥ 18 years
2. Confirmed haploidentical donor
3. Severe SCD phenotype who are at high risk for morbidity and mortality. Severe SCD is defined by at least one of the following:

i. Clinically significant neurologic event (stroke) or deficit lasting > 24 hours.

ii. History of ≥2 acute chest syndromes in a 2-year period preceding enrolment despite optimum treatment, e.g. with hydroxycarbamide (HC).

iii. History of ≥3 severe pain crises per year in a 2-year period preceding enrolment despite the institution of supportive care measures (e.g. optimum treatment with HC).

iv. Administration of regular transfusion therapy (=8 packed red blood transfusions per year for 1 year to prevent vaso-occlusive complications).

v. Patients assessed as requiring transfusion but with red cell allo-antibodies/very rare blood type, rendering it difficult to continue/commence chronic transfusion.

vi. Patients requiring HC/transfusion for treatment of SCD complications who cannot tolerate either therapy due to significant adverse reactions.

vii. Established end organ damage relating to SCD, including but not limited to progressive sickle vasculopathy and hepatopathy. End-organ sufficient for entry to this trial shall be ratified at the UK NHP.

d) Patients must be fit to proceed to Haploidentical SCT as defined below: i. Karnofsky score ≥60 ii. Cardiac function: LVEF ≥45% or shortening fraction ≥25% iii. Lung Function: FEV1, FVC and TLCO ≥50% iv. Renal function: EDTA GFR ≥40 ml/min/1.73m2 v. Hepatic function: ALT <x3 ULN and bilirubin <x2 the upper limit of normal, those with hyperbilirubinemia due to sickle related haemolysis will not be excluded. No radiological evidence of cirrhosis.

e) Written informed consent.

Exclusion Criteria:

1. Fully matched sibling donor.
2. Previous bone marrow transplant.
3. Pregnancy or breast feeding.
4. Participants able to conceive a child that are unprepared to use effective contraception.
5. Clinically significant donor specific HLA antibodies.
6. HIV infection or active Hepatitis B or C.
7. Uncontrolled infection including bacterial, fungal and viral.
8. Participation in another interventional trial in the last three months.
9. Pre-existing condition deemed to significantly increase the risk of Haploidentical SCT by the local Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Treatment failure or mortality | 24 months post-randomisation
  Treatment failure is defined as occurrence of vaso-occlusive crisis, or transfusion from 6 months post-randomisation.

SECONDARY OUTCOMES:
Health related quality of life | At 3, 6, 9, 12, 15, 18, 21 and 24 months post-randomisation
  Quality of life as measured by EQ-5D-5L
All cause mortality | 24 months post-randomisation
  Death by any cause
Sickle Cell Disease-related mortality (excluding transplant related complications) | 24 months post-randomisation
  Death due to any sickle cell disease related cause
Sickle type haemoglobin percentage (HbS%) | At 6, 12 and 24 months post-randomisation
  Sickle type haemoglobin as measured by haemoglobin electrophoresis
Sickle cell disease related complications | 24 months post-randomisation
  Defined as transfusion requirement, painful VOC, stroke, pulmonary hypertension
Haemoglobin levels, Reticulocyte count, LDH, Bilirubin | At 6, 12 and 24 months post-randomisation
Pulmonary Function | At 12 months and 24 months post-randomisation
  As measured by FEV1 %, FEV1/FVC ratio, TLCO %
Renal Function | At 6, 12 and 24 months post-randomisation
  As measured by urea, creatinine and eGFR
Iron overload | 24 months post-randomisation
  As measured by Ferritin and FerriScan (R2-MRI)
Cardiac function and pulmonary hypertension | At 12 and 24 months post-randomisation
  As measured by echocardiogram/TRV
Cerebrovascular progression | 24 months post-randomisation
  As measured by clinical stroke or evidence of progression on MRI/MRA
Evidence of hepatic progression | 24 months post-randomisation
  As measured by liver function (ALT, AST, ALP, GGT, Bilirubin) and FibroScan
Percentage of participants requiring opioid use for pain related to vaso-occlusive sickle related crisis | At 12 and 24 months post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Murtagh, Study Director — King's College Hospitals NHS Foundation Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided